CLINICAL TRIAL: NCT01787305
Title: Longitudinal Study of the Fecal Microbiome in Persistently Anti-β2 Glycoprotein-I Positive Individuals and Patients With Antiphospholipid Syndrome
Brief Title: Pilot Study of Gut Commensals in Antiphospholipid Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Hospital for Special Surgery, New York (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1210010962; U01AI101990 (NIH); R01AI118855-01 (NIH)
Record Dates: First submitted 2013-02-03; First posted 2013-02-08 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Antiphospholipid Syndrome (APS)
Keywords: microbiome; commensals; autoantibodies; autoreactive T cells
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole Blood Serum Stool DNA?
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to explore if certain commensals within the gut microbiota (the collection of all microbes that live inside the gut) correlate with autoantibodies in the autoimmune clotting disorder called antiphospholipid syndrome. The study hypothesis is that particular commensals induce the autoantibodies (immune molecules that bind to self structures) and thus correlate with the level of immune cells and antibodies that are self-reactive. Participants are patients with antiphospholipid syndrome and individuals who have tested positive on a prior blood test for anti-beta2-glycoprotein I antibodies or those that have tested negative for antiphospholipid antibodies in their blood, but had a clotting event or a health problem that puts them at risk to form blood clots.

DETAILED DESCRIPTION:
Antiphospholipid syndrome (APS) is an autoimmune disorder in which people are at risk to form blood clots. Having a positive antiphospholipid antibody (aPL) test does not mean the person has APS; but a small number of people do develop APS. These antibodies can also occur in otherwise healthy people. We believe certain bacteria in the gut may cause these antibodies to be produced.

Current treatments in APS target the blood clotting system and the goal is to prevent future blood clots. Many patients require this therapy for their entire life. If an persistent trigger can be found within the gut microbiota, it may help in developing other treatments. This study is being conducted at two centers, Yale University School of Medicine in New Haven, CT, and The Hospital for Special Surgery in Manhattan, New York. We expect to enroll a total of 40 subjects in this study at these study sites.

Visits will be as follows:

Visit 1: Initial screening visit: Review of medical records and questionnaire completion.

Visit 2 (one month after initial visit) & Visit 3 (2 months after initial visit): Questionnaire relating to any changes that may have taken place since recruitment. Brief physical examination by the study doctor.

Overall participation: Over a period of 8 weeks.

Sample Collection:

At each study visit, a sample of blood will be obtained (approximately 6.5 tablespoons of whole blood) via one needle stick.

A take-home stool sample collection kit will be provided. Stool samples will be obtained within 24 hours before or after blood collection and delivered (or mailed) to a study site. 2 kits will be provided at the initial visit, 1 kit will be provided at the follow up visit at month 1.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* One of the following groups below:

Group 1a: Persistently positive anti-β2GPI on Coumadin (n: 10) Group 1b: Persistently positive anti-β2GPI not on Coumadin (n: 10) Group 2a: Negative aPL on Coumadin (n: 10) Group 2b: Negative aPL not on Coumadin (n: 10) Persistently positive aβ2GPI will be defined as anti-β2GPI immunoglobulin G (IgG)/IgM/IgA ≥ 40 SGU/SMU at two separate time points at least 12 weeks apart.

Negative aPL will be defined as negative Lupus anticoagulant test, aCL IgG/IgM/IgA, and anti-β2GPI IgG/IgM/IgA within 12 months of the study entry.

Exclusion Criteria:

* Any autoimmune diseases including Rheumatoid Arthritis, Spondylarthropathy, Inflammatory Muscle Disease, and Sarcoidosis
* Steroid use greater than 10 mg/d prednisone or equivalent 30 days prior to enrollment
* Any immunosuppressive drug use within 3 months prior to screening (mycophenolate mofetil, azathioprine, methotrexate, leflunomide, rituximab, cyclophosphamide, intravenous immunoglobulin, plasmapheresis).
* Ongoing chronic infection (viral, bacterial or fungal) including known HIV, Hepatitis B/C
* Acute infection receiving any antibiotics within 30 days prior to screening
* Acute thrombosis within 2 days prior to screening
* Major gastrointestinal surgery less than 5 years prior to enrollment (with the exception of appendectomy)
* Any Gastrointestinal bleeding history
* Inflammatory Bowel Disease diagnosed by biopsy
* Celiac Disease diagnosed by biopsy
* Bulimia or anorexia nervosa
* Probiotics (greater than estimated 10^9 cfu or organisms per day) within 30 days prior to enrollment (with the exception of fermented beverages, milks or yogurts).
* Morbid obesity (BMI ≥ 40)
* Diabetes Mellitus Type I or II on medical therapy
* Malignancy within one year prior to screening (with the exception of non-metastatic squamous or basal cell skin carcinomas and cervical carcinoma if received curative surgical treatment)
* Known alcohol abuse
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Yale New Haven Hospital and affiliated outpatient clinics Hospital for Special Surgery and affiliated outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in autoantibody levels | Baseline
  Certain gut bacteria will correlate with anti-β2GPI autoantibody titers in anti-β2GPI-positive subjects that are lower or absent in aPL-negative subjects
Change in autoantibody levels | 4 weeks
  Certain gut bacteria will correlate with anti-β2GPI autoantibody titers in anti-β2GPI-positive subjects that are lower or absent in aPL-negative subjects
Change in autoantibody levels | 8 weeks
  Certain gut bacteria will correlate with anti-β2GPI autoantibody titers in anti-β2GPI-positive subjects that are lower or absent in aPL-negative subjects

SECONDARY OUTCOMES:
Change in autoreactive T cell frequencies | Baseline
  Certain gut bacteria will correlate with β2GPI-reactive CD4+ T-cells in anti-β2GPI-positive subjects that are lower or absent in aPL-negative subjects.
Change in autoreactive T cell frequencies | 4 weeks
  Certain gut bacteria will correlate with β2GPI-reactive CD4+ T-cells in anti-β2GPI-positive subjects that are lower or absent in aPL-negative subjects.
Change in autoreactive T cell frequencies | 8 weeks
  Certain gut bacteria will correlate with β2GPI-reactive CD4+ T-cells in anti-β2GPI-positive subjects that are lower or absent in aPL-negative subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Kriegel, MD PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine; Yale-New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Background] Ruff WE, Greiling TM, Kriegel MA. Host-microbiota interactions in immune-mediated diseases. Nat Rev Microbiol. 2020 Sep;18(9):521-538. doi: 10.1038/s41579-020-0367-2. Epub 2020 May 26. PMID 32457482
- [Result] Ruff WE, Dehner C, Kim WJ, Pagovich O, Aguiar CL, Yu AT, Roth AS, Vieira SM, Kriegel C, Adeniyi O, Mulla MJ, Abrahams VM, Kwok WW, Nussinov R, Erkan D, Goodman AL, Kriegel MA. Pathogenic Autoreactive T and B Cells Cross-React with Mimotopes Expressed by a Common Human Gut Commensal to Trigger Autoimmunity. Cell Host Microbe. 2019 Jul 10;26(1):100-113.e8. doi: 10.1016/j.chom.2019.05.003. Epub 2019 Jun 18. PMID 31227334